CLINICAL TRIAL: NCT01002040
Title: PCIRN Evaluation of Pandemic H1N12009 Influenza Vaccine in Adults With Human Immunodeficiency Virus Infection
Brief Title: Rapid Evaluation of Pandemic H1N1 Influenza Vaccine in Adults With HIV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H09-02820
Record Dates: First submitted 2009-10-23; First posted 2009-10-27 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: HIV Infections; H1N1 Influenza
Keywords: HIV; vaccine,; H1N1; influenza; H1N1 Influenza vaccine; Arepanrix; Pandemic; H1N1 2009 Influenza; HIV preventive vaccine
MeSH Terms: conditions — HIV Infections; Orthomyxoviridae Infections; Influenza, Human | interventions — arepanrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- One Dose Influenza vaccine (Active Comparator): Arepanrix H1N1 Influenza vaccine (one dose)
  Interventions: Biological: Arepanrix
- Two Doses Influenza vaccine (Active Comparator): Arepanrix H1N1 Influenza vaccine (2 doses, 3 weeks apart)
  Interventions: Biological: Arepanrix

INTERVENTIONS:
Biological: Arepanrix — Group A receives one dose of Arepanrix
  Arms: One Dose Influenza vaccine
Biological: Arepanrix — Group B receives 2 doses of Arepanrix 3 weeks apart
  Arms: Two Doses Influenza vaccine

SUMMARY:
The purpose of this study is to assess the safety and effectiveness (immune response) to a licensed H1N12009 influenza vaccine in HIV-infected adults. The study will enroll 150 adults (ages 20-59 years). Participants will be randomized into 2 groups and will receive either one dose or two doses of a licensed H1N1 vaccine. Study procedures include: medical history, blood samples and completing a memory aid. Participants will be involved in study related procedures for approximately 6 days.

DETAILED DESCRIPTION:
During the first wave of the H1N12009 pandemic in Canada, adults with immune deficiency were more likely to die with severe infections than were other Canadians. Of 76 deaths attributed to date to this new virus, 37% occurred in persons with immune system compromise. Adults with human immunodeficiency virus (HIV) infection constitute a significant proportion of the at-risk population with over 56,000 affected individuals. Most such individuals retain some capacity to respond to influenza vaccination. The dosing regimen for the pandemic vaccine will be based on limited studies in the general population, leaving open the question of whether HIV-infected persons can respond satisfactorily to the recommended dosing. Availability of an adjuvanted formulation of the pandemic vaccine may improve responsiveness but two doses may be required for the best possible response. Thus it would be optimal to evaluate the safety and immunogenicity of the pandemic vaccine among the earliest HIV-infected persons to receive it, to inform the subsequent vaccination of others.

The objectives of this study are three-fold:

1. To evaluate the safety and immunogenicity of H1N12009 influenza vaccine in a convenience sample of adults with HIV infection.
2. To compare immune responses of subjects randomized to receive either one or two doses of adjuvanted vaccine to identify the optimal regimen.
3. To complete this evaluation soon after the pandemic vaccine becomes available so as to inform the subsequent use of the vaccine in HIV-infected persons.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory-confirmed HIV
* Written informed consent
* Adults 20-59 years of age

Exclusion Criteria:

* Allergies to eggs, thimerosal or gentamicin sulphate
* Life-threatening reaction to previous Flu vaccine
* Bleeding disorder
* Pregnancy
* Receipt of blood or blood products in past 3 months
* Chronic illness
* Previous lab-confirmed H1N12009 infection
* Receipt of any non-study H1N12009 or Seasonal Influenza vaccine for 2009/10

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2010-02; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events (AEs) for days 0-6 after each vaccination | Day 7 and Day 21 post vaccination
Occurrence of serious adverse events (SAEs) and other significant health events up to 21 days after each vaccination | Day 7 and Day 21 post vaccination

SECONDARY OUTCOMES:
Immunogenicity: Comparison of baseline and post-immunization antibody titres | Day 21 post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: David Scheifele, MD, Principal Investigator — University of British Columbia; Curtis Cooper, MD, Study Director — University of Ottawa / Ottawa Hospital Research Institute,; Marina Klein, MD, Study Director — McGill University; Brian Ward, MD, Study Director — McGill University; Sharon Walmsley, MD, Study Director — University of Toronto; Allison McGeer, MD, Study Director — University of Toronto; David Hasse, MD, Study Director — Dalhousie University; Shelly McNeil, MD, Study Director — Dalhousie University
Locations (4):
- Canada (4):
  - Dalhousie University, Halifax, Nova Scotia
  - University of Ottawa / Ottawa Hospital Research Institute, Ottawa, Ontario
  - University of Toronto, Toronto, Ontario
  - McGill University, Montreal, Quebec

REFERENCES:
- [Derived] Cooper C, Klein M, Walmsley S, Haase D, MacKinnon-Cameron D, Marty K, Li Y, Smith B, Halperin S, Law B, Scheifele D; Phac Cihr Influenza Research Network. High-level immunogenicity is achieved vaccine with adjuvanted pandemic H1N1(2009) and improved with booster dosing in a randomized trial of HIV-infected adults. HIV Clin Trials. 2012 Jan-Feb;13(1):23-32. doi: 10.1310/hct1301-023. PMID 22306585